CLINICAL TRIAL: NCT06119438
Title: The Effect of Inhalation Aromatherapy on Pain and Anxiety Levels of The Patients Undergoing Prostate Biopsy: A Randomized Controlled Trial
Brief Title: Aromatherapy on Pain and Anxiety of the Patients Undergoing Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Barıs Saylam, Associate Proffesor, Mersin Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 375/2020
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Aromatherapy; Prostate Cancer; Anxiety
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: The study was designed as a placebo-controlled prospective double-blind study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Saline group (Active Comparator): Only saline solution was applied to the placebo group. The nebulizer was prepared and operated in the room where the prostate biopsy would be performed before the procedure. Patients were taken to the room 5 minutes before the procedure and the nebulizer was operated on during the procedure
  Interventions: Other: Aromatherapy
- Levander group (Active Comparator): Levander oil was added to the nebulizer at a rate of 2%. The nebulizer was prepared and operated in the room where the prostate biopsy would be performed before the procedure. Patients were taken to the room 5 minutes before the procedure and the nebulizer was operated during the procedure.
  Interventions: Other: Aromatherapy
- Frankincense group (Active Comparator): Frankincense oil was added to the nebulizer at a rate of 2%. Only saline solution was applied to the placebo group. The nebulizer was prepared and operated in the room where the prostate biopsy would be performed before the procedure. Patients were taken to the room 5 minutes before the procedure and the nebulizer was operated during the procedure.
  Interventions: Other: Aromatherapy

INTERVENTIONS:
Other: Aromatherapy — Aromatherapy is a TAT (Tapas Acupressure technique) method in which essential oils created from fragrant parts of plants are absorbed from the body and show their effects. The therapeutic, disease-relieving or preventive properties of essential oils are utilized

SUMMARY:
The study included 120 male patients who would undergo a prostate biopsy. Patients were divided into 3 groups as placebo group (n = 40), Levander group (N = 40), and Frankincense group (n = 40). Aromatherapy agents were added to the nebulizer at a rate of 2%. Only saline solution was applied to the placebo group. The nebulizer was prepared and operated in the room where the prostate biopsy would be performed before the procedure. Patients were taken to the room 5 minutes before the procedure and the nebulizer was operated during the procedure. The level of anxiety was evaluated by the State Anxiety Inventory (STAI-I). After the procedure, the patient was rested and were again filled out the STAI-1 form. After that, the data of all the patients involved in the study was compared.

DETAILED DESCRIPTION:
The study was conducted at Mersin University Medical Faculty Hospital Urology Department and Mersin City Training and Research Hospital Urology Department. The study was designed as a placebo-controlled prospective double-blind study. Approval was obtained from the Mersin University Ethics Committee for the study (13.05.2020, 375). All patients who participated were informed about the study and received written consent. The study included 120 male patients who would undergo a prostate biopsy. Exclusion criteria were identified as; patients with pain prior to the procedure (VAS value is non-zero), any respiratory disease (lung cancer, asthma, bronchitis, chronic obstructive pulmonary disease, etc.), patients using painkillers in the last 3 hours, patients who were disturbed by the smell of used essential oils and patients with a known allergy to used essential oils with a history of contact dermatitis against cosmetic odor. Patients with these characteristics were not included in the study. During transrectal ultrasound-guided prostate biopsy, periprostatic local anesthesia was routinely administered to all patients and is routinely performed in all prostate biopsies performed in the clinic. Patients have filled out STAI-2 (trait index) forms before the procedure. The STAI clearly distinguishes between the temporary situation of state anxiety and the more general and long-term quality of trait anxiety. The STAI index has 2 subheadings, STAI-1 (state index) and STAI-2 (trait index), with 40 questions. The scores of each subscale could range from a minimum of 20 to a maximum of 80. A score of 20-31 reflected mild anxiety, 32-42 below moderate anxiety, 43-53 above moderate anxiety, 54-64 relatively severe anxiety, and 65-75 severe anxiety. Patients were grouped and randomized according to the STAI-2 (trait index) scores.

Patients were divided into 3 groups placebo group (n = 40), Levander group (N = 40), and Frankincense group (n = 40). Aromatherapy agents were added to the nebulizer at a rate of 2%. Only saline solution was applied to the placebo group. The nebulizer was prepared and operated in the room where the prostate biopsy would be performed before the procedure. Patients were taken to the room 5 minutes before the procedure and the nebulizer was operated during the procedure. The level of anxiety was evaluated by the State Anxiety Inventory (STAI-I). The STAI-1 form was used to determine the transitory emotional state and anxiety level of the participants before and after the procedure. The interrogation procedures were carried out by an assistant doctor who had no knowledge about the study. After the procedure, the patient was rested and again filled out the STAI-1 form. After that, the data of all the patients involved in the study was compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing prostate biopsy

Exclusion Criteria:

* Patients with pain prior to the procedure (VAS value is non-zero),
* Patients with respiratory disease (lung cancer, asthma, bronchitis, chronic obstructive pulmonary disease, etc.),
* Patients using painkillers in the last 3 hours,
* Patients who were disturbed by the smell of used essential oils
* Patients with a known allergy to used essential oils with a history of contact dermatitis against cosmetic odor.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — patients underwent prostate biopsy
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
The STAI index | Immediately after the procedure.
  The STAI-1 form was used to determine the transitory emotional state and anxiety level of the participants before and after the procedure. The STAI index has 2 subheadings, STAI-1 (state index) and STAI-2 (trait index), with a total of 40 questions. The scores of each subscale could range from a minimum of 20 to a maximum of 80. Higher scores are positively correlated with higher levels of anxiety. A score of 20-31 reflected mild anxiety, 32-42 below moderate anxiety, 43-53 above moderate anxiety, 54-64 relatively severe anxiety, and 65-75 severe anxiety distinguishes between the temporary situation of state anxiety and the more general and long-term quality of trait anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Barış Saylam, Mersin, Mezitli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No